CLINICAL TRIAL: NCT02316145
Title: Internet-based Support and Coaching for Young Adults With Neuropsychiatric Disorders - A Pilot Study
Brief Title: Internet-based Coaching for Young Adults With Neuropsychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16611
Record Dates: First submitted 2011-12-20; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Tourette's Disorder
Keywords: ADHD; Autism spectrum condition; Tourette's disorder; Internet-based; chat; coach
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Tourette Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 'Habilitation (Internet-based support) (Other): Before the individual started with the internet-based support and coaching (IBSC), a meeting with the coach was compulsory to discuss what specific issues they were going to work with during the period of IBSC. The IBSC was offered at fixed times twice a week during an eight-week period. Two meetings between the individual and the coach were included. Between chat sessions the individuals and the coaches could get in touch using the programme's e-mail. The content of the support and coaching was individualised based on each individual's requirement. Once a fortnight a meeting was held with the head of the project and coaches. Issues regarding ongoing support and coaching were addressed.
  Interventions: Behavioral: Habilitation (Internet-based support and coaching)

INTERVENTIONS:
Behavioral: Habilitation (Internet-based support and coaching) — Support and coaching with therapist (psychologist or educational therapist) by using chat and e-mail

SUMMARY:
Purpose: To develop a model for internet-based support and coaching to young adults with neuropsychiatric disorders (NPD). To improve the individual's psychosocial functioning and his/her understanding of how he/she is functioning.

NPD comprise problems with social interaction, attention, impulse control and hyperactivity. The most common NPD diagnoses are ADHD (attention deficit hyperactivity disorder), autism spectrum condition (ASC) and Tourette's disorder (TD). In this study the investigators use Internet-based treatment for young adults with NPD.

Method: Support/coaching by using communication over the Internet (chat and e-mail) with individuals with NPD. Twice every week during 8 weeks, young adults with NPD are offered support and coaching over the Internet by psychologist/educational therapist with great experience from NPD. The individuals are assessed before and after treatment pertaining to quality of life, sense of coherence, self-esteem, depressive and anxiety symptoms, and parents' evaluation of the young adult's situation.

DETAILED DESCRIPTION:
Aims: To develop an internet-based support and coaching model for young people with autism spectrum disorder (ASD) and/or attention-deficit/hyperactivity disorder (ADHD), and to validate the model. Method: A user centred design was applied to develop a model for internet-based support and coaching, where individuals received eight-week support via internet (chat). The model was validated by ten individuals, 15 to 26 years of age, with ASD and/or ADHD. Self-report questionnaires (Sense of Coherence (SOC), the Rosenberg Self Esteem Scale, the Manchester Short Assessment of Quality of Life (MANSA), Montgomery Åsberg Depression Rating Scale (MADRS), and the Hospital Anxiety and Depression Scale (HAD)) were distributed before and after intervention. A structured interview regarding the quality of the model, the Patient perspective of Care and Rehabilitation process (POCR), was used after the intervention. Results: The validation showed significant improvement of SOC, self-esteem and subjective Quality of Life at follow-up and the majority perceived high fulfilment/importance on the POCR. Conclusions: The model can be an important complement to other interventions for young people with ASD and/or ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The individuals had to fulfill a diagnosis of ADHD, Tourette's disorder and/or an ASD (autistic disorder, Asperger's disorder or pervasive developmental disorder not otherwise specified (PDD NOS), according to the DSM-IV (APA, 1994).
* The inclusion age was between 15 and 26 years.

Exclusion Criteria:

* mental retardation,
* current psychosis,
* current major depression,
* current alcohol and/or substance abuse/dependence,
* severe dyslexia and/or severe psychosocial problems (e.g. criminality)

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
quality of life (QoL) | assessed at baseline; immediatelly after intervention and at 6-month follow-up
  The Manchester Short Assessment of Quality of Life (MANSA) is a 16-item scale that consists of four objective QoL questions and 12 questions pertaining to "life as a whole, job (or studies), financial situation, friendships, leisure activities, accommodation, personal safety, people that the person lives with, family and health".

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Wentz, MD, PhD, Study Chair — Child Neuropsychiatry Clinic